CLINICAL TRIAL: NCT03103659
Title: Optimization and Improvement of Care Course for 75 Years and Over Patient With Cancer and Living in Nursing Home on the Marseille Agglomeration
Acronym: ONCO-EHPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-48
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Cancer; Elderly
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly patient with cancer living in a nursing home (Experimental)
  Interventions: Other: personalised care plan

INTERVENTIONS:
Other: personalised care plan — Quality of life assessement in elderly cancer patients

SUMMARY:
According to data from the French National Cancer Institute (INCA), almost one third of the cancers were diagnosed in overs 75 years patients in France in 2008. The elderly patients management is an important part in oncology daily practice.

These last years, through the geriatric oncology development, collaboration between oncologists and geriatricians, the anti-cancer management and supportive care for elderly patients has evolved. The assessement of potential fragility helps to determine the cancers appropriate treatment plan.

Studies have shown that alterations in geriatric fields, found through Comprehensive Geriatric Assessment (CGA) are associated with poorer survival, increased risk of chemotherapy severe toxicity and autonomy loss.

Nursing home residents have often more frailties and functional problems than living at home elderly resulting in diagnostic and therapeutic cancer delay. In addition, nursing home residents must have appropriate treatment to preserve as much as possible their quality of life.

Transversal Onco-Geriatrics Unit (UTOG), Day Hospital (HDJ), External Geriatric Mobile Unit (EMGE) of the Internal Medicine, Geriatric and Therapeutic Department of the Marseille hospital propose to organize a personalized care course for nursing home residents with cancer to minimize the diagnostics delay, facilitate their management in oncology and maintain their quality of life.

Elderly patient with suspected cancer is oriented by EMGE to HDJ to realize an oncological and geriatric assessment. Patient would be supported by UTOG and would have access to technical platform.

According to his cancer and nursing home location, the nearest reference center would be offered.

Treatment or course of action (monitoring, palliative care …) would be decided in onco-geriatric multidisciplinary meeting (RCP) (organized by Onco-Geriatric Coordination Unit UCOG PACA west) and programmed and fast hospitalization would be organized in the reference center.

When returning in nursing homes, elderly patient would be revalued by EMGE to continue therapeutic management and personalized care plan. The aim of this management is to allow a shorter hospitalization and maintain the quality of life of frailty patient during cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with new diagnosis of cancer or follow-up breakdown or progression of the cancer disease

Exclusion Criteria:

* Elderly patients with cognitive impairment.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-27 (Estimated); Primary Completion 2018-04-27 (Estimated); Study Completion 2019-04-27 (Estimated)

PRIMARY OUTCOMES:
Time frame between diagnosis and access to oncologies care facilities | 6 months
  Number of days

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Couderc AL, Berbis J, Delalande G, Mugnier B, Courcier A, Bourriquen M, Rey D, Greillier L, Baciuchka M, Sudour P, Agnelli L, Nouguerede E, Fabries S, Villani P. Impact of care pathway for nursing home residents treated for cancer: ONCO-EHPAD study. Support Care Cancer. 2021 Jul;29(7):3933-3942. doi: 10.1007/s00520-020-05973-1. Epub 2021 Jan 3. PMID 33392770